CLINICAL TRIAL: NCT02493296
Title: The Effect of Surgery on Central Aortic Pressure & haEmodynamics Study
Acronym: ESCAPE
Status: Completed | Type: Observational
Sponsor: University of Leicester (Other)
Collaborators: British Heart Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 0066
Record Dates: First submitted 2015-07-06; First posted 2015-07-09 (Estimated); Last update posted 2020-01-30 (Actual); Status verified 2020-01

CONDITIONS: Abdominal Aortic Aneurysm; Pulse Wave Analysis; Risk
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Observational: The cohort will have their central aortic pressure, and carotid-femoral and brachio-femoral pulse-wave velocities measured. These measurements will take place pre-operatively, within a week of surgery, 6-weeks and 1-year post-operatively also. The surgery will be abdominal aortic aneurysm repair.
  Interventions: Other: This observational study will not entail an intervention.

INTERVENTIONS:
Other: This observational study will not entail an intervention. — This study will entail measurement of central aortic haemodynamics before and after (clinically indicated) abdominal aortic aneurysm repair

SUMMARY:
The present study will investigate the effect of artificially stiffening the aorta by means of an aortic stent on central aortic haemodynamics (CAH). This study will determine whether aortic stenting inadvertently adversely impacts on CAH, thereby providing the rational for subsequent therapeutic intervention to reduce the associated cardiovascular risk.

DETAILED DESCRIPTION:
Increased pulse pressure and pulse-wave velocity are recognized indices of arterial stiffness (Laurent, Boutouyrie, Asmar et al., 2001; Qiu, Winblad, Viitanen et al., 2003). An increased pulse pressure (indicative of increased central aortic pressure) is independently associated with an increased incidence of postoperative neurological and cardiac complications (Fontes, Aronson, Matthew et al., 2008). Pulse pressure has been identified as an independent predictor of cerebrovascular events after cardiac surgery (Benjo, Thompson, Fine et al., 2007). Moreover, many studies have demonstrated that pulse-wave velocity is an independent predictor of morbidity and mortality in a range of study populations (for a review see Vlachopoulos, Aznaouridis, Stefanadis, 2010). An increasing body of evidence suggests that brachial artery pressure, although representative, is not an accurate reflection of central aortic pressure. The Conduit Artery Function Evaluation study, for example, revealed that certain drugs preferentially reduce central aortic pressure, whilst having similar effects on brachial artery pressure. Moreover, in this study central aortic pulse pressure was demonstrated to be an independent predictor of clinical outcomes (Williams, Lacy, Thom et al., 2006). Other studies support the finding that markers of CAP are more closely related to surrogate measures of cardiovascular risk such as left ventricular mass (Haider, Larson, Franklin et al., 2003) and carotid intima-media thickness (Kostis, Davis, Cutler et al., 1997).

One inadvertent effect of stenting is the introduction of a semi rigid conduit into the circulation. This could potentially increase pulse wave velocity and adversely affect central aortic pressures and haemodynamics. The investigators thus aim to investigate the effect of aortic aneurysm of surgery on central aortic pressures and haemodynamics

ELIGIBILITY:
Inclusion Criteria:

* All participants undergoing abdominal aortic aneurysm repair, with non-atheromatous common carotid arteries.

Exclusion Criteria:

* Atheromatous carotid arteries

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All participants undergoing abdominal aortic aneurysm repair who are over 18, and are able to consent to the study.
Sampling Method: Non-Probability Sample
Enrollment: 146 (Actual)
Dates: Start 2010-10-07 (Actual); Primary Completion 2018-08-02 (Actual); Study Completion 2018-08-02 (Actual)

PRIMARY OUTCOMES:
Pulse wave velocity | One year

SECONDARY OUTCOMES:
Central aortic pressure | 1 Year

CONTACTS AND LOCATIONS:
Overall Officials: Vimal J Gokani, MBBS MRCS, Principal Investigator — University of Leicester
Locations (1):
- University of Leicester, Leicester, United Kingdom